CLINICAL TRIAL: NCT05386316
Title: Meeting Women Where They Are: The Maternal Health Multilevel Intervention for Racial Equity (MIRACLE) Project
Brief Title: The Maternal Health Multilevel Intervention for Racial Equity (MIRACLE) Project
Acronym: MIRACLE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Corewell Health West (Other); Hurley Medical Center (Other); Ascension Health (Industry)
Responsible Party: Principal Investigator, Jennifer E. Johnson, C. S. Mott Endowed Professor of Public Health, Michigan State University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01MD016003 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-23 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Maternal Morbidity and Mortality; Health Disparities
Keywords: maternal mortality; maternal health; maternal health services; African American; health disparity; healthcare disparities
MeSH Terms: conditions — Maternal Death | interventions — Mortality; erucylphosphocholine

STUDY DESIGN:
Intervention Model Description: Individuals who live in the intervention counties at the time of birth will be assigned to the intervention condition. Individuals who live in control counties at the time of birth are assigned to the control condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data include Medicaid claims and birth and death records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention counties (Experimental): Birthing persons who live in Kent County or Genesee County, Michigan, USA at the time of delivery.
  Interventions: Other: Multilevel intervention for racial disparities in severe maternal morbidity and mortality; Other: Standard Enhanced Prenatal Care (EPC) services
- Control counties (Active Comparator): Birthing persons who live in the other Michigan, USA counties at the time of delivery.
  Interventions: Other: Standard Enhanced Prenatal Care (EPC) services

INTERVENTIONS:
Other: Multilevel intervention for racial disparities in severe maternal morbidity and mortality — In addition to standard enhance prenatal care (EPC) services, the following will be offered.
  Community level. We will make EPC services (i.e., MIHP and Healthy Start) available via telehealth with flexible hours to women who are eligible for Healthy Start (primarily minority women) who decline traditional (i.e., home visiting) services.
  Provider/practice level. We will provide actionable maternal health-focused anti-racism training to health system administrators, physicians, residents, midwives, nurses, front desk staff, schedulers, public health officers, EPC staff, doulas, WIC staff, and lactation consultants.
  System level. Counties will implement equity focused community care maternal safety bundles. Community care is care provided by outpatient, EPC, community-based organizations, and linkages between hospital care and these settings.
  Arms: Intervention counties
Other: Standard Enhanced Prenatal Care (EPC) services — Pregnant women in comparison counties will receive whatever EPC services (MIHP and/or Healthy Start) they naturalistically choose to receive.
  Maternal Infant Health Program (MIHP). All women in Michigan who are Medicaid insured are eligible for MIHP. MIHP offers monthly home visiting and care coordination to supplements regular care during pregnancy and up to 12 months post birth. MIHP offers care coordination; risk assessment; individual care plan; evidence-based interventions; transportation; education; and referrals.
  Healthy Start. Health Start is a federally funded program for minority women that offers more intensive EPC services delivered by race/ethnicity matched community health workers. Community health workers offer peer support; resilience and problem solving; risk assessment; facilitating provider-client communication; collaborative care; system navigation, including transition from prenatal care to postnatal primary care; and supportive referrals.

SUMMARY:
This community-partnered study will scale a community, provider, and system-level implementation intervention to reduce African American maternal morbidity and mortality disparities in two Michigan counties (Genesee and Kent). This project will test the intervention using data from Medicaid insured women who deliver in Michigan from 2016-2019 and 2022-2025 (approximately 540,000 births, including 162,000 births to African American women).

DETAILED DESCRIPTION:
Maternal morbidity and mortality in the US are critical problems of public health significance. US maternal mortality rates are the highest among high-income countries. In addition, severe maternal morbidity (SMM; "unexpected outcomes of labor and delivery that result in significant short- or long-term consequences to a woman's health"1), affects around 60,000 US women every year. Such life-threatening complications affect mothers, children, families, and communities, and cost billions of dollars per year.

These challenges disproportionately affect African American (AA) women. AA women are three to four times more likely to die of pregnancy related complications than non-Hispanic white (NHW) women and have twice the rates of SMM.2,3 Inequities occur at many levels. These include the community level, in which the built environment and working multiple jobs while managing family obligations can make it difficult for AA women to access even enhanced prenatal and postnatal care (EPC) programs designed for them. At the provider/practice level, implicit and explicit biases and the structures and practices reflecting them contribute to inadequate quality of care for AA women, reduce the acceptability of treatment, and contribute to racial disparities in maternal morbidity and mortality. At the system level, health systems serving AA women are less likely to offer high-quality care, and quality initiatives that to do not directly target disparities often have little or no effect on disparities.

This proposal will test the effectiveness and cost-effectiveness of a multilevel intervention to address AA-NHW maternal morbidity and mortality disparities in two Michigan counties: Genesee County (which includes Flint) and Kent County (which includes Grand Rapids). Interventions at each level were developed or co-developed by our partners in these counties, who include AA women residents and community leaders, EPC staff (including Community Health Workers), and physician/health system representatives.

Community level (improving accessibility) intervention. This project will expand access to EPC services using telehealth and flexible scheduling (e.g. outside business hours). EPC programs (such as Healthy Start and statewide home visiting programs) provide care coordination, promote healthy behaviors, provide health education and social support, and address social determinants of health. These programs, some using race-matched Community Health Workers, improve maternal and infant health, including reducing mortality, especially for AA. Despite being designed for minority women, 60% of eligible AA women in Michigan do not enroll in EPC services. The investigators found that 50% of minority women who declined EPC services said they would participate if a tele-health option was available. This project will provide this option to improve access to these important services.

Provider/practice level (improving acceptability) intervention. This project will address provider and health system implicit and explicit bias and corresponding structures and practices and make this learning actionable using daylong experiential trainings. Trainings will include didactics, reflection, discussion, windshield tours, and brainstorming ways to tailor trainees' settings to better hear, respect, and meet the needs of perinatal AA women. Training will include everyone from physicians to front desk staff and will take place in small groups (10-20) with additional opportunities for the larger community to come together to brainstorm and plan responses.

System level (improving quality) intervention. This project will deploy community care patient safety bundles targeting maternal health disparities throughout the intervention counties. Community care is defined as care provided by outpatient, EPC, and community-based organizations. Kent County is the lead of 5 pilot communities in the national Alliance for Innovation on Maternal Health Community Care Initiative (AIM-CCI) to develop and implement non-hospital focused maternal safety bundles. The bundles provide care guidelines to address disparities in preventable maternal mortality and SMM. As part of this project, Genesee County will implement the bundles in partnership with Kent County, providing the final level of our multilevel intervention.

The study sample will include all Medicaid insured women observed during pregnancy, at birth, and/or up to 1 year postpartum, who deliver in Michigan from 2016-2019 and 2021-2024 (~540,000 births, including ~162,000 births to AA women). Investigators will test the effects of the multilevel intervention using a quasi-experimental difference-in-difference with propensity scores approach to compare pre (2016-2019) to post (2022-2025) changes in outcomes among Medicaid women in the two intervention counties with similar women in other counties. Measures will be taken from a pre-existing linked dataset that includes Medicaid claims, death records, birth records, and EPC program data. The specific aims are to:

1. Assess the effectiveness of the multilevel intervention on the following outcomes:

   1. AA SMM and pregnancy-related mortality (up to 1-year postpartum; overall & relative to NHW women)
   2. AA non-severe maternal morbidity (overall & relative to NHW women)
2. Test improved service utilization (enrollment in EPC, more outpatient visits, fewer emergency department [ED] visits during pregnancy and postpartum) and non-severe maternal morbidity (overall & relative to NHW women) as mechanisms of the effect of the multilevel intervention on SMM
3. Evaluate the cost-effectiveness of the multilevel intervention

AA women face addressable disparities in maternal morbidity and mortality. This trial, among the first to evaluate a multilevel intervention to address population-level AA SMM, will help build the evidence-base to address them. The study will also provide information about cost-effectiveness needed to drive policy decisions and information about mechanisms of intervention effects needed to drive the science forward. Achieving these aims will deter-mine whether this intervention could be scaled widely to reduce AA SMM and pregnancy-related mortality.

ELIGIBILITY:
Inclusion Criteria: Resided in intervention county at time of delivery. -

Exclusion Criteria: None.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All birthing persons, regardless of self-identified gender.
Enrollment: 540000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
severe maternal morbidity | Pregnancy through 12 months postpartum
  We will assess severe maternal morbidity (SMM, as defined by CDC and ACOG)4 using CDC's list of 21 SMM indicators based on ICD-10 diagnosis and procedure codes.60 The binary overall SMM indicator will be coded 1 if any SMM will be identified during a woman's pregnancy, delivery, and up to 12 months postpartum using Medicaid claims and 0 otherwise.
severe maternal morbidity + pregnancy-related mortality | Pregnancy through 12 months postpartum
  An indicator representing yes/no any SMM and/or pregnancy-related mortality

SECONDARY OUTCOMES:
non-severe maternal morbidity | pregnancy through 12 months postpartum
  Measurement of "non-severe" maternal morbidity (NSMM), is taken from the WHO's Maternal Morbidity Working Group (MMWG).61-64 Most NSMM are measurable using ICD-10 diagnostic and procedure codes63,65 To capture multimorbidity in our sample, the overall NSMM indicator will be the sum of WHO-delineated NSMM diagnoses and procedures63,65 identified in a woman's Medicaid claims during pregnancy and up to 1 year postpartum. We will also assess the following WHO-defined subcategories: (1) number of direct NSMM diagnoses and procedures (e.g., delivery complications, hypertensive disorders of pregnancy, obstetric hemorrhage, pregnancy-related infections);63 (2) number of indirect NSMM diagnoses and procedures (e.g. endocrine, nutritional, and metabolic diseases; mental disorders); and (3) number co-incidental NSMM (e.g. partner violence, sexual assault) diagnoses and procedures.63
enrollment in enhanced prenatal care | pregnancy through 12 months postpartum
  Binary indicator reflecting yes/no enrollment in MIHP and/or Health Start
outpatient visits | pregnancy through 12 months postpartum
  Number of outpatient pregnancy and postpartum visits (higher is better)
emergency department visits | pregnancy through 12 months postpartum
  Number of emergency department visits (lower is better)
cost-effectiveness | pregnancy through 12 months postpartum
  The primary outcome used for cost-effectiveness analyses will be SMM. Prevented SMM will be monetized using Medicaid claims data by calculating the difference between Medicaid delivery expenditures between women with SMM and without SMM using our own claims data and prior estimates.6 Secondary cost-effectiveness measures will be maternal mortality and NSMM. The value of a statistical life,66 currently around $10 million, will be used to monetize prevented maternal deaths. For NSMM, we will calculate intervention costs per point of NSMM score reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Johnson, PhD, Principal Investigator — Michigan State University; Cristian Meghea, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We can share fidelity data generated by the project, but we cannot share routinely collected MDHHS warehouse data (i.e., Medicaid claims, birth and death records) accessed by this project because it will not be generated by the project. Access to MDHHS data requires a data use agreement and a specific request to MDHHS from each research team. Study results will be shared widely with community, practice, and policy partners using a variety of approaches, as well as through standard academic channels.

REFERENCES:
- [Derived] Johnson JE, Roman L, Key KD, Meulen MV, Raffo JE, Luo Z, Margerison CE, Olomu A, Johnson-Lawrence V, White JM, Meghea C. Study protocol: The Maternal Health Multilevel Intervention for Racial Equity (Maternal Health MIRACLE) Project. Contemp Clin Trials. 2022 Sep;120:106894. doi: 10.1016/j.cct.2022.106894. Epub 2022 Aug 24. PMID 36028193
- See also: Study web page — https://obgyn.msu.edu/research/the-miracle-study
- See also: News article — https://publichealth.msu.edu/news-items/research/255-nih-grant-to-address-maternal-morbidity-and-mortality-disparities